CLINICAL TRIAL: NCT01644942
Title: Identification in Obese Patients of the Mechanisms Involved in Intramuscular Lipid Accumulation.
Brief Title: Identification in Obese Patients of the Mechanism Involved in Intramuscular Lipid Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 8193
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Obesity; Insulin Resistance; Hyperlipidemia
Keywords: Obese; insulin sensitive; insulin resistant; myotubes; lipid accumulation
MeSH Terms: conditions — Obesity; Insulin Resistance; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin sensitive patients (Other)
  Interventions: Other: Lipid accumulation analysis
- Insulin resistant patients (Other)
  Interventions: Other: Lipid accumulation analysis

INTERVENTIONS:
Other: Lipid accumulation analysis — The lipid accumulation will be assessed with muscular biopsies.

SUMMARY:
The study aims to determine in obese patients the implication of intramuscular lipid accumulation in relation with insulin resistance and defect in lipid oxidation.

DETAILED DESCRIPTION:
Obese insulin sensitive and obese insulin resistant patients undergo a glucose tolerance test, indirect calorimetry during exercise and muscular biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with a Body Mass Index (BMI) between 30 and 40 kg/m2
* Patients who do not practice physical exercise (Voorips index < 9)
* Age between 40 and 70 years- Male gender
* Fast blood glucose <1,10 g/l and no hypoglycemic treatment
* Signed informed consent
* Social security affiliation
* Absence of anti VIH, anti hepatitis C antibodies, and HBS antigen
* Normal biological tests
* Non smoking persons

Exclusion Criteria:

* Patients who refuse the anti-VIH, anti-hepatitis C antibodies, and HBS antigens tests
* Patients treated by anticoagulant, b blockers, lipopenic, or anti-inflammatory.
* Patients with a contraindication to muscular exercise (retinopathy, coronaropathy, nephropathy) and to muscular biopsy
* Allergy to local anaesthetic

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
lipid accumulation in skeletal muscle | 1 month

SECONDARY OUTCOMES:
lipid accumulation in myotubes from obese patients | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Montpellier, Montpellier, France